CLINICAL TRIAL: NCT04838210
Title: Elevating Voices, Addressing Depression, Toxic Stress and Equity in Group Prenatal Care
Acronym: EleVATE GC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202103142
Record Dates: First submitted 2021-03-18; First posted 2021-04-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related; Perinatal Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Prenatal Care (Experimental): Group prenatal care model
  Interventions: Behavioral: EleVATE Group Care
- Individual Prenatal Care (Active Comparator): Individual prenatal care
  Interventions: Behavioral: Individual Prenatal Care

INTERVENTIONS:
Behavioral: EleVATE Group Care — 10-session (2 hours per session) group prenatal care model following the prenatal visit schedule recommended by ACOG. In addition to pregnancy and infant-care related content, the EleVATE GC curriculum includes behavioral health strategies that can be used to manage depression and labor pain and navigate the daily frustrations and stress of life. Groups are facilitated by an obstetric clinician.
  Arms: Group Prenatal Care
Behavioral: Individual Prenatal Care — The dominant model of prenatal care in the United States, consisting of one-on-one encounters between a patient and obstetric clinician. Patients are seen for 10-15 mins every 4 weeks until 28 weeks gestation, every 2 weeks until 37 weeks or more by provider discretion), and weekly until delivery. Visits focus on routine screening tests and prenatal care.
  Arms: Individual Prenatal Care

SUMMARY:
This study will provide high-quality, representative data on the capacity of Elevating Voices, Addressing Depression, Toxic Stress and Equity in Group Prenatal Care (EleVATE GC) to reduce perinatal depression, preterm birth, and low birthweight in African-American women. If findings from this study indicate that EleVATE GC is feasible and effective, this model could be implemented nationwide to help achieve mental and obstetric health parity for low-income women of color in the United States.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* ≤18 weeks' gestation
* Established prenatal care at EleVATE site
* High-risk for postpartum depression by ≥1 risk factor (personal/family history, baseline EPDS≥10, low-income, 13-19 years old, single, history of physical/sexual abuse, unplanned/undesired pregnancy, history of pregnancy loss)
* Ability to attend group prenatal visits at specified days/times
* Willingness to be randomized
* Ability to give informed consent
* Any patient that has received prenatal care in a group setting previously

Exclusion Criteria:

* Multiple gestation
* Major fetal anomaly
* Serious medical co-morbidity/psychiatric illness necessitating more care than can be safely provided in group setting
* Serious medical co-morbidity necessitating more care than can be safely provided in group setting

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Depression | Baseline visit
  Major Depression (Edinburgh Postnatal Depression Scale Score, range: 0-30, higher scores are a worse outcome)
Perinatal Depression | 28-40 week visit
  Major Depression (Edinburgh Postnatal Depression Scale Score, range: 0-30, higher scores are a worse outcome)
Perinatal Depression | 4-12 weeks Postpartum
  Major Depression (Edinburgh Postnatal Depression Scale Score, range: 0-30, higher scores are a worse outcome)

SECONDARY OUTCOMES:
Preterm Birth | Delivery
  Delivery at <37 weeks gestation
Small for Gestational Age | Delivery
  Birthweight <10th percentile on the Alexander growth curve
Perceived Stress | Baseline visit
  Perceived Stress Scale Total Scores, range: 0-40, higher scores are a worse outcome
Perceived Stress | 28-40 week
  Perceived Stress Scale Total Scores, range: 0-40, higher scores are a worse outcome
Perceived Stress | 4-12 weeks Postpartum
  Perceived Stress Scale Total Scores, range: 0-40, higher scores are a worse outcome
Anxiety | Baseline visit
  PROMIS Short Form Anxiety 8a T-Score, range: 37.1-83.1, higher scores are a worse outcome
Anxiety | 28-40 week visit
  PROMIS Short Form Anxiety 8a T-Score, range: 37.1-83.1, higher scores are a worse outcome
Anxiety | 4-12 weeks Postpartum
  PROMIS Short Form Anxiety 8a T-Score, range: 37.1-83.1, higher scores are a worse outcome
Post-Traumatic Stress Disorder (PTSD) | Baseline Visit
  PTSD Checklist for DSM-V Total Symptom Severity Score, range 0-80, higher scores are a worse outcome
Social Support | Baseline visit
  PROMIS Bank 2.0 Social Support (emotional support, instrumental support, informational support, and social isolation domains) T-Scores, range 23.7-76.9, higher scores are better outcomes for emotional support, instrumental support and informational support, higher scores are worse outcomes for social isolation
Social Support | 28-40 week visit
  PROMIS Bank 2.0 Social Support (emotional support, instrumental support, informational support, and social isolation domains) T-Scores, range 23.7-76.9, higher scores are better outcomes for emotional support, instrumental support and informational support, higher scores are worse outcomes for social isolation
Social Support | 4-12 weeks Postpartum
  PROMIS Bank 2.0 Social Support (emotional support, instrumental support, informational support, and social isolation domains) T-Scores, range 23.7-76.9, higher scores are better outcomes for emotional support, instrumental support and informational support, higher scores are worse outcomes for social isolation
Race-Related Stress | Baseline visit
  Index of Race Related Stress-Brief Version Total Score, range 0-22, higher scores are worse outcomes
Maternal Attachment (Antenatal) | Baseline visit
  Maternal Antenatal Attachment Scale Total Score, range 19-95, higher scores are better outcomes
Maternal Attachment (Antenatal) | 28-40 week visit
  Maternal Antenatal Attachment Scale Total Score, range 19-95, higher scores are better outcomes
Maternal Attachment (Postnatal) | 4-12 Weeks Postpartum
  Maternal Postnatal Attachment Scale Total Score, range 19-95, higher scores are better outcomes

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Missouri-Kansas City/Truman Health Centers-Kansas City, Kansas City, Missouri
  - Affinia Healthcare, St Louis, Missouri
  - Family Care Health Centers, St Louis, Missouri
  - CareSTL Health, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes